CLINICAL TRIAL: NCT05011045
Title: Neurocognitive Outcomes After Whole Brain Radiation Therapy for Hematologic Malignancies
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA18-0791; PA18-0791 (Other: M D Anderson Cancer Center); NCI-2021-08429 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Central Nervous System Lymphoma; Hematopoietic and Lymphoid Cell Neoplasm; Leukemia; Lymphoma; Plasma Cell Myeloma; Secondary Central Nervous System Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma | interventions — Magnetic Resonance Spectroscopy; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (neurocognitive assessment, questionnaires, MRI): Patients undergo neurocognitive function assessments, complete questionnaires over 8-10 minutes and undergo standard of care MRI at baseline (within 4 weeks before the first day of WBRT), 2, 6, 12 months after RT completion, then annually for 5 years.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Neurocognitive Assessment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Neurocognitive Assessment — Undergo neurocognitive function assessment
Other: Quality-of-Life Assessment — Complete questionnaires
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study assesses neurocognitive outcomes after receiving radiation therapy to the brain (whole brain radiation therapy) in patients with blood cancers (hematologic malignancies). This may help researchers learn more about the effects of whole brain radiation therapy on memory and thinking in patients with blood cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Record patients' cognitive outcomes after whole-brain radiation therapy (WBRT) for hematologic malignancies using standard-of-care neurocognitive function testing.

SECONDARY OBJECTIVES:

I. Assess patients' quality-of-life after WBRT for hematologic malignancies, based on a validated questionnaire.

II. Explore magnetic resonance imaging (MRI) changes in the brain after WBRT for hematologic malignancies, based on standard-of-care imaging studies.

III. Study the role of Memantine in patients' cognitive outcomes during and after WBRT for hematologic malignancies, based on standard-of-care use, utilizing standard-of-care neurocognitive function testing.

OUTLINE:

Patients undergo neurocognitive function assessments, complete questionnaires over 8-10 minutes and undergo standard of care MRI at baseline (within 4 weeks before the first day of WBRT), 2, 6, 12 months after RT completion, then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Treatment with radiation therapy to the brain for a hematologic malignancy (ex. primary central nervous system lymphoma [PCNSL], secondary central nervous system lymphoma [SCNSL], leukemia, myeloma)
* Proficient and capable of completing tests in English
* Patients with claustrophobia are eligible if the claustrophobia is managed with medication
* Patients with cognitively-impairment are eligible if the impairment is managed with medication
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiation therapy to the brain for a hematologic malignancies
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive outcomes | Up to 5 years
  Neurocognitive failure will be defined as the first cognitive failure on 2 or more of the following tests: the Hopkins Verbal Learning Test Revised Total Recall, Delayed Recall and Delayed Recognition; the Controlled Oral Word Association; and the Trail Making Test Part A or B. The rate of neurocognitive failure and its 95% confidence interval (CI) will be calculated. The cumulative incidence approach may be used to estimate the median time to neurocognitive failure to account for the competing risk of death. May use the Aalen-Johansen estimator of the cumulative incidence function.

SECONDARY OUTCOMES:
Quality-of-life | Up to 5 years
  Assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Core 30/Brain Neoplasm 20. The rates of improvement and worsening will be calculated. The rate of deterioration will be calculated. Also, Wilcoxon signed rank test or paired t-test will be used to compare the scores between baseline and after radiation at 2 months.
Magnetic resonance imaging (MRI) changes | Baseline up to 5 years
  Will explore radiographic changes on standard-of-care MRI scans that are suggestive of radiation toxicity. Radiographic changes will be considered in the context of radiation treatment plans. Correlation of radiographic changes with radiation dose will be performed for hypothesis generation. Spearman correlation coefficient may be used to assess the correlation between radiographic changes and radiation dose.
Role of medications indicated to improve memory and cognitive function | Up to 5 years
  Neurocognitive outcomes at different time points will be summarized using descriptive statistics. Changes overtime on neurocognitive outcomes may be analyzed using generalized linear models for the repeated measures. May compare the neurocognitive outcomes of the patients to a similar cohort of patients that were not treated with Memantine or other medications indicated to improve memory and cognitive function (example the RT arm of RTOG 1114). Will amend the protocol to include the details on which cohort of patients to be compared to, variables to be used for matching the two patient cohorts, and method to be used for matching once decided to proceed with the comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina S Dabaja, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States